CLINICAL TRIAL: NCT00663923
Title: Comparison of Cross-cylinder and Conventional PRK for Laser Correction of Astigmatism: A Randomized Clinical Trial.
Brief Title: Comparison of Cross-cylinder and Conventional Photorefractive Keratectomy(PRK) in Correcting Medium-high Astigmatism
Acronym: PRK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 86-43
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2011-12-30 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Astigmatism
Keywords: Excimer Laser; photorefractive keratectomy; astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cross-cylinder (Experimental): In this technique the laser is programmed with the axis and amount of cylinder,so that the steepest meridian is flattened with central cylindrical ablation and the flattest meridian steepens with paracentral ablation
  Interventions: Procedure: photorefractive keratectomy (PRK)
- single (Active Comparator): In this technique ,cylinder is treated only on one meridian by performing an elliptical ablation to to flatten the steeper meridian to match the flatter meridian.
  Interventions: Procedure: photorefractive keratectomy (PRK)

INTERVENTIONS:
Procedure: photorefractive keratectomy (PRK) — comparison of PRK by cross-cylinder approach in one eye and conventional (single) method in the other eye for laser correction of astigmatism
  Other Names: photoastigmatic keratectomy

SUMMARY:
The purpose of this study is to determine whether cross-cylinder approach is more effective than routine method in laser correction of astigmatism.

DETAILED DESCRIPTION:
Both eyes of 50 patients(100 eyes) with medium-high compound myopic astigmatism and inclusion criteria,will be treated by photorefractive keratectomy (PRK) using excimer laser.It breaks chemical bonds within corneal stroma.It's wavelength is 193 nm that is in the ultraviolets range with high energy and very low tissue penetrance. The right or left eye of every patient would be allocated randomly to one of the study groups using RandList 1.1. In spite of recent advances in excimer laser machines and surgical techniques,correction of astigmatism is not more successful compared to myopia. In this study we will compare two methods of laser correction of astigmatism regarding to visual acuity,residual error and aberrations.

ELIGIBILITY:
Inclusion Criteria:

* >20 years of age
* refractive stability for at least one year
* regular and symmetric astigmatism of >1.5 diopters

Exclusion Criteria:

* corneal thickness<470 microns
* keratoconus or suspected keratoconus
* active ocular disease and systemic collagen disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Sedghipoor, MD, Study Director — Ophthalmology Department, Tabriz University of medical Sciences
Locations (1):
- Nikookari eye hospital, Tabriz, East Azerbaijan Province, Iran

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both eyes of Fifty patients with medium-high compound myopic astigmatism(1.5- 5 D) were enrolled in a prospective randomized study between sep 2007 and sep 2008 at Nikookari eye hospital and Mehr eye center
Pre-assignment Details: All enrolled patients having inclusion criteria accepted both available techniques for correction of astigmatism.
Groups:
- Photorefractivekeratectomy(PRK): Right or left eye of 50 patients was randomly enrolled(data provided in this module refer to 100 eyes of 50 participants)to undergo PRK by cross-cylinder or conventional(single) approach using Excimer laser.In cross-cylinder method , half of the cylinder is treated along the steepest meridian and the other half is ablated along the flattest meridian .in single method,the steepest meridian is treated by elliptical ablation to match the flattest meridian.
Period: Overall Study
Arm/Group | Photorefractivekeratectomy(PRK)
Started | 50
Completed | 48
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Photorefractive Keratectomy( PRK): Right or left eye of 50 patients was randomly enrolled(data provided in this module refer to100 eyes of 50 participants)to undergo PRK by cross-cylinder or conventional(single) approach using Excimer laser.In cross-cylinder method , half of the cylinder is treated along the steepest meridian and the other half is ablated along the flattest meridian .In single method the steepest meridian is treated by elliptical ablation to match the flattest meridian.
Arm/Group | Photorefractive Keratectomy( PRK)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.46 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants] — one eye of 39 females and 11 males underwent PRK by cross-cylinder approach and the other eye underwent PRK by single method
  Participants
    Female | 39
    Male | 11
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 50
Target induced astigmatism(TIA) [Mean (Standard Deviation); unit: Diopter] — It is vector of astigmatic change intended to be induced by the surgery. Participant population was the same as baseline participants. It was measured by refraction(using autorefractor) and vector analysis(using special software).Diopter is a unit of measurement of the optical power of any refracting surface ,which is reciprocal of the focal length measured in meters.
  Diopter | 1.86 (0.60)
astigmatism [Mean (Standard Deviation); unit: diopter] — In compound myopic astigmatism the meridians of maximum and minimum power are both too strong.So both line images fall short of the retina.Participant population was the same as baseline population.
  It was measured by refraction(using autorefractor).Diopter is a unit of measurement of the optical power of any refracting surface ,which is reciprocal of the focal length measured in meters.
  diopter | -2.49 (0.83)
corrected distance visual acuity [Mean (Standard Deviation); unit: logMAR] — Corrected VA is attained after correction of refractive errors using lenses of varying powers .the data are the LogMAR values calculated from the snellen chart using the visual acuity conversion chart(the units would be LogMAR).Any patient with better vision can see the smallest letters at 20 feet(20/20=0.00 LogMAR).Higher LogMAR values represent worse outcome.LogMAR(logarithmic minimum angle of resolution)notation has gained widespread use in statistical calculations.
  logMAR | 0.06 (0.11)
high order aberration [Mean (Standard Deviation); unit: micron] — Although lower- order aberrations decrease after laser vision correction,higher -order aberrations may increase after conventional PRK or lasik.Higher-order aberration is Composed of delicate irregularities within the cornea not correctable by spectacles.It is measured using aberrometer.In this study OPD scan was used for aberrometry which is one of the methods of wavefront analysis.Participant population was the same as baseline population.
  micron | 0.36 (0.10)
Spherical equivalent [Mean (Standard Deviation); unit: Diopter] — Average of the maximum and minimum powers,which equals the sphere power plus half the cylinder power.Participant population was the same as baseline population.
  It was measured by refraction(using autorefractor).Diopter is a unit of measurement of the optical power of any refracting surface ,which is reciprocal of the focal length measured in meters.
  Diopter | -5.19 (2.47)
uncorrected distance visual acuity [Mean (Standard Deviation); unit: log MAR] — Uncorrected VA is attained before correction of refractive errors .the data are the LogMAR values calculated from the snellen chart using the visual acuity conversion chart(the units would be LogMAR).Any patient with better vision can see the smallest letters at 20 feet(20/20=0.00 LogMAR).Higher LogMAR values represent worse outcome.Log MAR(logarithmic minimum angle of resolution)notation has gained widespread use in statistical calculations.
  log MAR | 1.11 (0.36)

OUTCOME MEASURES:

1. Primary Outcome: Correction of Astigmatism
Description: It shows the result of correction of astigmatism .In compound myopic astigmatism the meridians of maximum and minimum power are both too strong.So both line images fall short of the retina.It is measured by refraction(using autorefractor).Diopter is a unit of measurement of the optical power of any refracting surface ,which is reciprocal of the focal length measured in meters.
Time Frame: six months after surgery
Population: The sample size was determined by the one proportion formula where power = 0.8, d=0.02 , p= 0.5(primary outcome) and type I error probability associated with this test of null hypothesis is 0.05.
  The analysis was per protocol
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Groups:
- Cross-cylinder PRK: Right or left eye of 50 patients was randomly enrolled(data provided in this module refer to 50 eyes of 50 participants)to undergo PRK by cross-cylinder approach using Excimer laser.In this method , half of the cylinder is treated along the steepest meridian and the other half is ablated along the flattest meridian .
- Single PRK: Right or left eye of 50 patients was randomly enrolled(data provided in this module refer to 50 eyes of 50 participants)to undergo PRK by single approach using Excimer laser.In this method ,the steepest meridian is treated by elliptical ablation to match the flattest meridian.
Arm/Group | Cross-cylinder PRK | Single PRK
Number analyzed (Participants) | 48 | 48
Number analyzed (eyes) | 48 | 48
diopter | -0.54 (0.43) | -0.59 (0.33)
Statistical Analysis 1: Comparison: Cross-cylinder PRK vs Single PRK; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — two - tailed p value <0.05 were considered statistically significant; in this study degrees of freedom is sample size - 1; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-.62 to -.001], Standard Deviation .10

2. Secondary Outcome: Higher Order Aberrations
Description: Although lower- order aberrations decrease after laser vision correction,higher -order aberrations may increase after conventional PRK or LASIK(Laser in situ keratomileusis).Higher-order aberration is Composed of delicate irregularities within the cornea not correctable by spectacles.It is measured using aberrometer.In this study OPD scan was used that is one of the methods of wavefront analysis .
Time Frame: six months postoperative
Population: the analysis was per protocol.
Measure: Mean (Standard Deviation); unit: micron
Units Other Than Participants: eyes
Arm/Group | Cross-cylinder PRK | Single PRK
Number analyzed (Participants) | 42 | 42
Number analyzed (eyes) | 42 | 42
micron | 0.51 (0.21) | 0.51 (0.20)

3. Secondary Outcome: Corrected Distance Visual Acuity(CDVA)
Description: CDVA is attained after correction of refractive errors using lenses of varying powers .the data are the LogMAR values calculated from the snellen chart using the visual acuity conversion chart(the units would be LogMAR).Any patient with better vision can see the smallest letters at 20 feet(20/20=0.00 LogMAR).Higher LogMAR values represent worse outcome.Log MAR(logarithmic minimum angle of resolution)notation ,has gained widespread use in statistical calculations.
Time Frame: six months
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Cross-cylinder PRK | Single PRK
Number analyzed (Participants) | 48 | 48
Number analyzed (eyes) | 48 | 48
LogMAR | 0.02 (0.02) | 0.03 (0.03)

4. Secondary Outcome: Uncorrected Distance Visual Acuity (UCDVA)
Description: UCDVA is attained without correction of refractive errors .the data are the LogMAR values calculated from the snellen chart using the visual acuity conversion chart( the units would be LogMAR).Any patient with better vision can see the smallest letters at 20 feet(20/20=0.00 LogMAR).Higher LogMAR values represent worse outcome.Log MAR(logarithmic minimum angle of resolution)notation ,has gained widespread use in statistical calculations.
Time Frame: six months
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Arm/Group | Cross-cylinder PRK | Single PRK
Number analyzed (Participants) | 48 | 48
Number analyzed (eyes) | 48 | 48
LogMAR | 0.08 (0.15) | 0.10 (0.16)

5. Secondary Outcome: Surgically Induced Astigmatism
Description: It is the vector of the astigmatic change actually induced by the surgery.Participant population was the same as baseline participants.
  It was measured by refraction(using autorefractor) and vector analysis(using special software).Diopter is a unit of measurement of the optical power of any refracting surface ,which is reciprocal of the focal length measured in meters
Time Frame: six months after surgery
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Cross-cylinder PRK | Single PRK
Number analyzed (Participants) | 48 | 48
Diopter | 1.98 (0.57) | 1.51 (0.43)

ADVERSE EVENTS:
Arm/Group | Cross-cylinder PRK | Single PRK
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No